CLINICAL TRIAL: NCT06771648
Title: A Prospective, Single-arm, Open-label, Post-market Clinical Follow-up Investigation to Verify Performance and Safety of Daxxin Psoriasis Shampoo When Used for Treatment of Moderate Scalp Psoriasis
Brief Title: Daxxin Psoriasis Shampoo PMCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daxxin AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAX_001
Record Dates: First submitted 2024-12-19; First posted 2025-01-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Scalp Psoriasis
Keywords: scalp psoriasis; shampoo; PMCF; Daxxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scalp psoriasis (Experimental): Subjects with the diagnosis of moderate scalp psoriasis
  Interventions: Device: Daxxin Psoriasis Shampoo

INTERVENTIONS:
Device: Daxxin Psoriasis Shampoo — Daxxin Psoriasis Shampoo at least 3 times a week and at most once a day as per instructions for use

SUMMARY:
The goal of this clinical investigation is to verify the performance and safety of the CE-marked Daxxin Psoriasis Shampoo to treat scalp psoriasis. Forty-one subjects with moderate scalp psoriasis are planned to be recruited at one site in Sweden. Subjects will be asked to use the shampoo between 3 and 7 times a week, as per the instructions for use from the manufacturer, for a period of 6 weeks.

DETAILED DESCRIPTION:
Investigational device: Daxxin Psoriasis Shampoo, Basic UDI-DI: 733116220030

Intended use: Daxxin Psoriasis Shampoo is designed to alleviate symptoms related to scalp psoriasis, such as itchiness, redness, flaking, and scratch marks

Overall design:

This is a prospective, single-arm, open-label, post-market clinical follow-up investigation designed to verify performance and safety of Daxxin Psoriasis Shampoo when used by subjects with scalp psoriasis in need of treatment. The outcome will be evaluated and incorporated in the product specific clinical evaluation report (CER) and serve as a base for continuous investigations.

Following approval from the ethical committee (EC), 41 subjects with the diagnosis of moderate scalp psoriasis will be recruited at sites in Sweden. The subjects should only use Daxxin Psoriasis Shampoo and no other shampoo during the study period.

The overall duration of the investigation is estimated to 8 months, including a 6-months recruitment period. Expected duration of each subject's participation is 6 weeks with 4 visits at site. The investigation will be considered complete when the last subject has completed the last visit.

Description of Medical Procedure:

Daxxin Psoriasis Shampoo should be used at least 3 times a week and at most once a day (7 times per week). Daxxin Psoriasis Shampoo should be used according to the instruction for use (IFU), and it is important to leave the shampoo in the hair and scalp for 2-5 minutes after massaging a generous foam.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old
2. Clinical diagnosis of moderate scalp psoriasis assessed by Psoriasis Scalp Severity Index (PSSI, moderate = 3-10)
3. At least a score of 1 grade for each symptom erythema, induration and desquamation
4. Subject is willing and able to use Daxxin Psoriasis Shampoo as directed, comply with investigation instructions, and commit to all follow-up visits for the duration of the investigation, as judged by the Investigator
5. Subject agrees to refrain from using other treatments for scalp psoriasis during the clinical investigation
6. Subject is willing and able to provide written informed consent

Exclusion Criteria:

1. Known allergy or sensitivity to any component of the device
2. Use of psoriasis shampoo 2 weeks prior to enrolment
3. Use of other psoriasis scalp treatment i.e., Betnovate that could affect the study result within 4 weeks prior to enrolment
4. Use of systemic and/or biological treatment for psoriasis
5. Subject has a history of psoriasis unresponsive to topical treatments
6. Subject is pregnant, lactating at time of enrolment, or is planning to become pregnant during the study
7. Subjects with any other condition that, as judged by the investigator, may make investigation procedures inappropriate
8. Subject with alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
PSSI score reduction at day 42 | From Day 0 (enrollment) to Day 42 after enrollment of each subject
  Percentage of subjects with reduction of at least 1-grade in the PSSI (Psoriasis Scalp Severity Index) score, at Visit 4 (Day 42) compared to Day 0 (baseline).

SECONDARY OUTCOMES:
PSSI score reduction at Days 14 and 28 | From Day 0 (enrollment) to Day 28 after enrollment of each subject
  Percentage of subjects with reduction of at least 1-grade in the PSSI score, at Visit 2 (Day 14) and Visit 3 (Day 28) compared to Day 0 (baseline).
DLQI | From Day 0 (enrollment) to Day 42 after enrollment of each subject
  Change in Quality of Life assessed with Dermatology Life Quality Index Scale (DLQI) from baseline (Day 0) to Visit 2 (Day 14), to Visit 3 (Day 28), Visit 4 (Day 42)
Scratch mark grades | From Day 0 (enrollment) to Day 42 after enrollment of each subject
  Change in scratch mark grades from baseline (Day 0) to Visit 2 (Day 14), to Visit 3 (Day 28), and to Visit 4 (Day 42)
Itching | From Day 0 (enrollment) to Day 42 after enrollment of each subject
  Change in subject reported itching, assessed with scalp-specific itch NRS, from baseline (Day 0) to end of treatment Visit 4 (Day 42) including weekly reports
Subject reported symptoms | From Day 0 (enrollment) to Day 42 after enrollment of each subject
  Change in subject reported symptoms (itching, redness, and flaking) using Likert scale from baseline (Day 0) to Visit 2 (Day 14), to Visit 3 (Day 28), and to Visit 4 (Day 42)
Subject satisfaction | Day 42 after enrollment of each subject
  To evaluate subject satisfaction after using Daxxin Psoriasis Shampoo, measured with a Likert scale at Visit 4 (Day 42).
Device usability | Day 42 after enrollment of each subject
  To evaluate device usability as measured by a Likert scale at Visit 4 (Day 42).
Safety | From the enrollment of the first subject to the last visit of the last subject, which is planned to correspond to a 8-month period
  Incidence of AEs, adverse device effects (ADEs), serious adverse events (SAEs), serious adverse device effects (SADEs), and device deficiencies (DDs) throughout the clinical investigation

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - CTC, Mölndal
  - Enheten för kliniska studier, University Hospital Region Örebro, Örebro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crowley J. Scalp psoriasis: an overview of the disease and available therapies. J Drugs Dermatol. 2010 Aug;9(8):912-8. PMID 20684141
- [Background] Mosca M, Hong J, Hadeler E, Brownstone N, Bhutani T, Liao W. Scalp Psoriasis: A Literature Review of Effective Therapies and Updated Recommendations for Practical Management. Dermatol Ther (Heidelb). 2021 Jun;11(3):769-797. doi: 10.1007/s13555-021-00521-z. Epub 2021 Apr 24. PMID 33893995
- [Background] Papadimitriou I, Bakirtzi K, Katoulis A, Ioannides D. Scalp Psoriasis and Biologic Agents: A Review. Skin Appendage Disord. 2021 Nov;7(6):439-448. doi: 10.1159/000517806. Epub 2021 Aug 3. PMID 34901174
- [Background] Blakely K, Gooderham M. Management of scalp psoriasis: current perspectives. Psoriasis (Auckl). 2016 Mar 29;6:33-40. doi: 10.2147/PTT.S85330. eCollection 2016. PMID 29387592